CLINICAL TRIAL: NCT06919107
Title: Use of Advanced Footwear Technology in Federated Athletes. An Ambispective Observational Study
Brief Title: Advanced Footwear Technology in Federated Athletes
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Ruben Cuesta Barriuso, Principal Investigator, University of Oviedo
Other Study IDs: ATL-foot
Record Dates: First submitted 2025-03-25; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Athlete Foot
Keywords: Disease; Athletics; Advanced Footwear Technology; Risk; Secondary Prevention; Physiotherapy
MeSH Terms: conditions — Tinea Pedis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Athletes using advanced footwear technology: Athletes competing in events longer than 800 meters, federated in the Athletics Federation of the Principality of Asturias and using shoes with Advanced Footwear Technology. Data will be collected on the number of injuries (muscle and tendon), lower limb injuries in the last 3 athletic seasons, as well as age, sex, weekly training load with and without AFT, weekly training frequency, completion of a complementary toning program and foot size
  Interventions: Other: Survey of athletes

INTERVENTIONS:
Other: Survey of athletes — Data will be collected on the number of injuries (muscle and tendon), lower limb injuries in the last 3 athletic seasons, as well as age, sex, weekly training load with and without AFT, weekly training frequency, completion of a complementary toning program and foot size.

SUMMARY:
Background. Athletics is one of the sports modalities with the greatest growth in the number of federative licenses in our country. In the last five years, the use of footwear with Advanced Footwear Technology (AFT) has become widespread in order to increase athletic performance.

Objective. To analyze the risk of injury in athletes using Advanced Footwear Technology as well as the sporting, sociodemographic and anthropometric variables that influence this risk.

Method. Ambispective cohort study. Ninety-five athletes competing in events longer than 800 meters will be recruited. The primary variable will be the number of injuries, muscular and tendon, of lower limbs in the last 3 athletic seasons. Secondary and modifying variables will be: age, sex, weekly training load with and without AFT, weekly training frequency, completion of a complementary toning program and foot size. Potential confounding variables will be body mass index, main training surface and commercial footwear models used. The analysis will calculate the risk of injury in these athletes and assess the influence of confounders and trend analysis on the primary variable, stratified by potential confounders.

Expected results. To calculate the risk of injury as a function of sport, sociodemographic and anthropometric variables. Identify

ELIGIBILITY:
Inclusion Criteria:

* Athletes competing in events longer than 800 meters; iii) athletes who have not undergone previous musculoskeletal surgery in the seasons under study.
* Federated in the Federación de Atletismo del Principado de Asturias (Asturias Athletics Federation).
* Athletes who have not undergone previous musculoskeletal surgery in the seasons under study.
* Who were federated at least one year before the study period.

Exclusion Criteria:

* Athletes who do not use AFT devices.
* Athletes with a muscle or tendon injury at the time of the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Federated athletes competing in events over 800 meters in the Principality of Asturias.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the number of muscle and tendon injuries recorded by athletes in the lower limbs | Screening visit
  Number of lower limb muscle and tendon injuries during the last 3 athletic seasons

SECONDARY OUTCOMES:
Assessment of age | Screening visit
  Measurement of age (measured in years completed, by requesting the date of birth to calculate this value).
Assessment of gender | Screening visit
  Measurement of gender (measured with a dichotomous variable: female / male)
Assessment of the weekly training load, using AFT or not | Screening visit
  Measurement of weekly training load with and without AFT (measured in kilometers traveled)
Assessment of weekly training frequency | Screening visit
  Measurement of weekly training frequency (measured in hours).
Assessment of the implementation of a complementary strengthening program | Screening visit
  Measurement of the implementation of a complementary strengthening program (measured with a dichotomous variable: yes/no).
Assessment of the size of athletes' feet | Screening visit
  Measurement of foot size (measured in international units)

OTHER OUTCOMES:
Assessment of body mass index | Screening visit
  Measurement of body mass index (measured as kg/m2). This variable will be considered as a possible confounding variable
Assessment of the main training surface | Screening visit
  Measurement of the main training surface (response options: asphalt, dirt, track and tartan). This variable will be considered as a possible confounding variable
Assessment of commercial footwear models used by athletes | Screening visit
  Measurement of commercial footwear models used (response options: Nike ZoomX Vaporfly NEXT%, Nike ZoomX Alphafly NEXT%, Adidas Adizero Adios Pro, Asics Metaspeed Sky, New Balance Fuelcell SuperComp Elite, Saucony Endorphin Pro, Puma Deviate Nitro Elite, and HOKA Rocket X). This variable will be considered as a possible confounding variable
Assessment of athletes' weight | Screening visit
  Assessment of athletes' weight, measured in kg.
Assessment of the height of the athletes | Screening visit
  Assessment of the height of the athletes, measured in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Study Director — Universidad de Oviedo
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided